CLINICAL TRIAL: NCT00871702
Title: Infusion of Genetically Modified T Cells: A Pilot Study of Tracking and Toxicity
Brief Title: Infusion of Genetically Modified T Cell for Post Transplant Patients With Relapsed Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0744 / 201103095
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Multiple Myeloma
Keywords: Leukemia; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Donor lymphocyte infusion (Experimental): CD34-TK75 transduced T lymphocytes from donors matched at a 5/6 or 6/6 antigen level at a dose of 1.0 x 105 cells/kg recipient weight.
  Interventions: Genetic: CD34-TK75 transduced donor lymphocytes; Radiation: Sub Study - 18 FHBG PET/CT Scans

INTERVENTIONS:
Genetic: CD34-TK75 transduced donor lymphocytes
Radiation: Sub Study - 18 FHBG PET/CT Scans — Three 18 FHBG PET/CT Scans will be performed first one at pre-DLI infusion, second 14 days post-DLI infusion and third 30 days post-DLI infusion - patients #3 - #8

SUMMARY:
Primary Objective:

* To determine if there is significant toxicity associated with the administration of CD34-TK75 transduced donor lymphocytes after allogeneic BMT for relapsed hematologic malignancies

Secondary Objectives:

* To determine if the patient develops any evidence of anti-leukemic effect from the administration of CD34-TK75 transduced donor lymphocytes
* To determine if ganciclovir administration to patients who develop Graft versus Host Disease (GVHD)results in clinical improvement after infusions of CD34-TK75 transduced lymphocytes.

Sub-Study Objective

The primary purpose is to perform PET imaging of CD34-TK transduced allogeneic donor T cells in patients who have relapsed hematologic malignancies after allogeneic hematopoietic stem cell transplantation (SCT). At this time the limited amount of cGMP quality virus produced by the NGVL will likely permit the imaging of only 3 patients. Consequently our current objective will be to establish that the TK-expressing cells can be detected by 18FHBG-PET in patient organs relevant for performing additional studies that are currently in the planning stages and for which we are working to produce additional virus.

The ultimate objective will be to use the TK substrate 18FHBG to locate the donor T cells within the recipient as they exert anti-leukemic effects, and the T cells can then be eliminated in response to in vivo administration of ganciclovir, before morbidity and mortality from GvHD occurs. We will use the imaging strategy to define patterns of T cell trafficking in humans pre and post-DLI infusion, and to determine where the cells reside while they mediate GVL in contrast to GvHD. We expect to obtain in vivo PET imaging markers predictive of GvHD before clinical symptoms occur.

DETAILED DESCRIPTION:
This is a phase I study of to determine the safety of the administration of lymphocytes, collected from the bone marrow donor. Donor lymphocytes are often administered in the case of a relapsed cancer after allogeneic bone marrow transplantation, in the hope to reduce the amount or size of the relapsed cancer. In this study, we will look for a decrease of the size of the relapsed cancer.

By inserting genetic material (DNA) into the cells (lymphocytes) collected from the donor, these cells will be genetically modified and made very sensitive to the killing effects of a drug called ganciclovir, routinely used in the clinic after bone marrow transplantation to treat virus infections in transplant patients.

This research study is to determine, if administration of the drug ganciclovir to the recipient, after intravenous infusion of the genetically modified cells (lymphocytes) into the recipient, will reduce or even eliminate a life threatening complication of allogeneic transplantation, called graft versus host disease (GvHD). The drug ganciclovir will kill the infused genetically modified donor cells (lymphocytes) so they cannot cause GvHD.

In summary, the overall purpose of this research study is to determine, if administration of a seven day course of the drug ganciclovir to the donor lymphocyte recipient will either decrease the severity of GvHD, or will decrease the number of cases with life-threatening GvHD after donor lymphocyte infusions.

This study will also determine if insertion of a small piece of DNA (a small piece of genetic material), makes these donor lymphocytes opened up and sensitive to the killing effects of the drug ganciclovir, but at the same time does not harm the lymphocytes' ability to reduce the amount or size of the cancer in the recipient. The DNA to be inserted into the donor lymphocytes is transported into these cells by a type of virus called "retrovirus vector". This retrovirus vector is made so the virus cannot divide (cannot make more of itself), and cannot make cells or the recipient sick. Retroviruses do, however, allow for the gene (DNA) they are carrying, to be permanently inserted into the genetic material of the donor lymphocytes. Therefore, this inserted DNA will persist in the donor lymphocytes for the life of the lymphocytes.

Finally, this study will also determine if the administration of genetically manipulated donor lymphocytes is well tolerated.

Sub Study

The goal of this subproject is to see if an imaging procedure called 18FHBG-PET/CT can help us see if the lymphocytes you received have gone to the sites in the body where the anti-cancer effects are taking place.

ELIGIBILITY:
Inclusion Criteria for Patient:

* Patients must be prior recipients of allogeneic BMT (matched 6/6 or 5/6 according to the National Marrow Donor Program) for any hematologic malignancy. Eligible patients would include those with leukemia, non Hodgkins Lymphoma, Hodgkins Disease, myelodysplastic syndrome and multiple myeloma.
* Patients must have laboratory, histologic, or cytogenetic evidence of disease relapse after allogeneic BMT.
* Patients may not have received prior therapy with transduced or non-transduced donor lymphocytes.
* Patients ≥ 18 years of age.
* The minimum number of transduced and purified lymphocytes from the same donor of donated cells for allogeneic transplant is is 1x105 per kg for all patients.
* Expected survival of patient is at least 4 weeks.
* Required baseline organ function within 14 days prior to study entry:

  * Renal function with creatinine less than 5 mg/dl.
  * Liver function with SGOT, SGPT and alkaline phosphatase ≤ 4 times the upper limit of institutional normal.
  * Bilirubin ≤ 5.0 mg/dl.
* Patient must have signed the informed consent prior to entry and express willingness to meet all the expected requirements of the protocol for the duration of the study.
* ECOG Performance Status ≤ 2
* All patients must agree to a repeat bone marrow, liver, gastro-intestinal or skin biopsies dependent on clinical course.
* Women of child bearing potential must have a negative pregnancy test (ß-HCG ) within 7 days of study entry.
* In addition patients # 3 to 8:

  * Must have consented to participation in HRPO 09-0744, "Infusion of Genetically Modified T cells: A Pilot I Study of Tracking and Toxicity
  * Must be willing to undergo 18FHBG-PET/CT-imaging
  * Must be able to tolerate 45-60 minutes of imaging at each imaging timepoint.
  * Women of child bearing potential must have an additional negative high sensitivity pregnancy test (20mlU ß-HCG /ml urine as administered in the Center for Clinical Imaging Research, Mallinckrodt Institute of Radiology, Washington University) prior to each imaging session (i.e. at days 10-16 and days 27-33).

Inclusion Criteria for Donor:

* Must be the original donor for the allogeneic bone marrow transplant patient.
* No underlying conditions which would contra-indicate apheresis.
* Must have signed the informed consent and express willingness to meet all the expected requirements stated in the protocol for the duration of the study.
* Must be eligible according to Washington University "Guidelines for Eligibility of Normal Donors"
* Donors ≥ 18 years of age.
* Female donors of childbearing potential must have a confirmed negative pregnancy test.

Exclusion Criteria for Patient:

* Patients receiving immunosuppression (cyclosporin, FK506, prednisone, cellcept, methylprednisolone) for GvHD or other reasons at the time of lymphocyte infusion.
* Patients must not have evidence of active CMV or other active viral infection requiring antiviral therapy. A culture or PCR of blood for CMV must be negative for enrollment.
* Pregnant or lactating females.Note that a second and third high sensitivity pregnancy test (20mlU ß-HCG /ml urine as administered in the Center for Clinical Imaging Research, Mallinckrodt Institute of Radiology, Washington University) are required prior to each imaging session (i.e. at days 10-16 and days 27-33 for patients #3 to 8).
* Uncontrolled infection: Any uncontrolled viral, bacterial, or fungal infection.
* HIV infection.
* Acute medical problems such as ischemic heart or lung disease.
* Patients with any underlying conditions which would contra-indicate therapy with study treatment (or allergies to reagents used in this study).
* Patients who have received atgam, campath [alemtuzumab] or daclizumab within 4 weeks of DLI.
* Patients receiving investigational drugs or treatments within 30 days of enrollment.
* Patients with tetracycline, penicillin, or streptomycin sensitivity.
* Patients with signs of acute GVHD as defined by the International Bone Marrow Transplant Registry (IBMTR) Severity Index for Acute Graft versus Host Disease (Rowlings, et al., Brit. J. Haematol. 97:855-64 [1997]). In addition patients may be excluded at the discretion of the treating physician.
* In addition for patients # 3 to 8 who will be imaged , exclude:

  * Patients who are claustrophobic.
  * Patients who are unable to tolerate 30-45 minutes of imaging.

Exclusion Criteria for Donor:

-Pregnant female donors

Concomitant Medication and Treatment:

-The principal investigator or a designated co-investigator at the respective institution must approve use of chemotherapeutic, antiviral or immunosuppressive medications.

Medications and Treatments Not Allowed:

-No other forms of chemotherapy will be administered after cell infusion during the treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To determine if there is significant toxicity associated with the administration of CD34-TK75 transduced donor lymphocytes after allogeneic BMT for relapsed hematologic malignancies | Day 0 through Day 100
  Occurrence of grade 3-5 toxicity
  72 hour infusional toxicity
  Acute GVHD
Perform PET imaging to allow us to locate the donor T cells within the recipient as they exert anti-leukemic effects, and the T cells can then be eliminated in response to administration of ganciclovir, before morbidity and mortality from GvHD occurs | Baseline, Day 14, and Day 30
To determine if there is significant toxicity associated with the administration of CD34-TK75 transduced donor lymphocytes after allogeneic BMT for relapsed hematologic malignancies | Day 100 - Year 15
  Occurrence of grade 3-5 toxicity

SECONDARY OUTCOMES:
To determine if the patient develops any evidence of anti-leukemic effect from the administration of CD34-TK75 transduced donor lymphocytes | 100 days
To determine if GCV administration to patients who develop GvHD results in clinical improvement after infusions of CD34-TK75 transduced lymphocytes. | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: John F. DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Rettig MP, Ritchey JK, Meyerrose TE, Haug JS, DiPersio JF. Transduction and selection of human T cells with novel CD34/thymidine kinase chimeric suicide genes for the treatment of graft-versus-host disease. Mol Ther. 2003 Jul;8(1):29-41. doi: 10.1016/s1525-0016(03)00142-4. PMID 12842426
- [Background] Rettig MP, Ritchey JK, Prior JL, Haug JS, Piwnica-Worms D, DiPersio JF. Kinetics of in vivo elimination of suicide gene-expressing T cells affects engraftment, graft-versus-host disease, and graft-versus-leukemia after allogeneic bone marrow transplantation. J Immunol. 2004 Sep 15;173(6):3620-30. doi: 10.4049/jimmunol.173.6.3620. PMID 15356106
- [Background] Drobyski WR, Keever CA, Roth MS, Koethe S, Hanson G, McFadden P, Gottschall JL, Ash RC, van Tuinen P, Horowitz MM, et al. Salvage immunotherapy using donor leukocyte infusions as treatment for relapsed chronic myelogenous leukemia after allogeneic bone marrow transplantation: efficacy and toxicity of a defined T-cell dose. Blood. 1993 Oct 15;82(8):2310-8. PMID 8400284
- [Background] Moolten FL. Tumor chemosensitivity conferred by inserted herpes thymidine kinase genes: paradigm for a prospective cancer control strategy. Cancer Res. 1986 Oct;46(10):5276-81. PMID 3019523
- [Background] Moolten FL, Wells JM. Curability of tumors bearing herpes thymidine kinase genes transferred by retroviral vectors. J Natl Cancer Inst. 1990 Feb 21;82(4):297-300. doi: 10.1093/jnci/82.4.297. PMID 2299679
- [Background] Miller AD, Buttimore C. Redesign of retrovirus packaging cell lines to avoid recombination leading to helper virus production. Mol Cell Biol. 1986 Aug;6(8):2895-902. doi: 10.1128/mcb.6.8.2895-2902.1986. PMID 3785217
- [Background] Kasid A, Morecki S, Aebersold P, Cornetta K, Culver K, Freeman S, Director E, Lotze MT, Blaese RM, Anderson WF, et al. Human gene transfer: characterization of human tumor-infiltrating lymphocytes as vehicles for retroviral-mediated gene transfer in man. Proc Natl Acad Sci U S A. 1990 Jan;87(1):473-7. doi: 10.1073/pnas.87.1.473. PMID 2404283
- [Background] Tiberghien P, Reynolds CW, Keller J, Spence S, Deschaseaux M, Certoux JM, Contassot E, Murphy WJ, Lyons R, Chiang Y, et al. Ganciclovir treatment of herpes simplex thymidine kinase-transduced primary T lymphocytes: an approach for specific in vivo donor T-cell depletion after bone marrow transplantation? Blood. 1994 Aug 15;84(4):1333-41. PMID 8049449
- [Background] Bordignon C, Bonini C, Verzeletti S, Nobili N, Maggioni D, Traversari C, Giavazzi R, Servida P, Zappone E, Benazzi E, et al. Transfer of the HSV-tk gene into donor peripheral blood lymphocytes for in vivo modulation of donor anti-tumor immunity after allogeneic bone marrow transplantation. Hum Gene Ther. 1995 Jun;6(6):813-9. doi: 10.1089/hum.1995.6.6-813. PMID 7548281
- [Background] Tiberghien P, Ferrand C, Lioure B, Milpied N, Angonin R, Deconinck E, Certoux JM, Robinet E, Saas P, Petracca B, Juttner C, Reynolds CW, Longo DL, Herve P, Cahn JY. Administration of herpes simplex-thymidine kinase-expressing donor T cells with a T-cell-depleted allogeneic marrow graft. Blood. 2001 Jan 1;97(1):63-72. doi: 10.1182/blood.v97.1.63. PMID 11133743
- [Background] Black ME, Newcomb TG, Wilson HM, Loeb LA. Creation of drug-specific herpes simplex virus type 1 thymidine kinase mutants for gene therapy. Proc Natl Acad Sci U S A. 1996 Apr 16;93(8):3525-9. doi: 10.1073/pnas.93.8.3525. PMID 8622970
- [Background] Szer J, Grigg AP, Phillips GL, Sheridan WP. Donor leucocyte infusions after chemotherapy for patients relapsing with acute leukaemia following allogeneic BMT. Bone Marrow Transplant. 1993 Feb;11(2):109-11. PMID 8435660
- [Background] Bar BM, Schattenberg A, Mensink EJ, Geurts Van Kessel A, Smetsers TF, Knops GH, Linders EH, De Witte T. Donor leukocyte infusions for chronic myeloid leukemia relapsed after allogeneic bone marrow transplantation. J Clin Oncol. 1993 Mar;11(3):513-9. doi: 10.1200/JCO.1993.11.3.513. PMID 8445426
- [Background] Kolb HJ, de Witte T, Mittermuller J, et al. (1993) Graft-versus-leukemia effect of donor buffy coat transfusions on recurrent leukemia after marrow transplantation. Blood 82: 214A
- [Background] Kolb HJ, Schattenberg A, Goldman JM, Hertenstein B, Jacobsen N, Arcese W, Ljungman P, Ferrant A, Verdonck L, Niederwieser D, van Rhee F, Mittermueller J, de Witte T, Holler E, Ansari H; European Group for Blood and Marrow Transplantation Working Party Chronic Leukemia. Graft-versus-leukemia effect of donor lymphocyte transfusions in marrow grafted patients. Blood. 1995 Sep 1;86(5):2041-50. PMID 7655033
- [Background] Blaese RM, Culver KW, Miller AD, Carter CS, Fleisher T, Clerici M, Shearer G, Chang L, Chiang Y, Tolstoshev P, Greenblatt JJ, Rosenberg SA, Klein H, Berger M, Mullen CA, Ramsey WJ, Muul L, Morgan RA, Anderson WF. T lymphocyte-directed gene therapy for ADA- SCID: initial trial results after 4 years. Science. 1995 Oct 20;270(5235):475-80. doi: 10.1126/science.270.5235.475. PMID 7570001
- [Background] Marktel S, Magnani Z, Ciceri F, Cazzaniga S, Riddell SR, Traversari C, Bordignon C, Bonini C. Immunologic potential of donor lymphocytes expressing a suicide gene for early immune reconstitution after hematopoietic T-cell-depleted stem cell transplantation. Blood. 2003 Feb 15;101(4):1290-8. doi: 10.1182/blood-2002-08-2351. Epub 2002 Oct 3. PMID 12393508
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu